CLINICAL TRIAL: NCT06439719
Title: Differences in Plaque Composition Evaluated Through Coronary Tomography in Subjects With Type 2 Diabetes With and Without Microvascular Complications
Brief Title: Plaque Composition in T2DM With and Without Microvascular Complications
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6561
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- T2DM with microvascular complications: T2DM with microvascular complications
  Interventions: Procedure: Blood sample collection
- T2DM without microvascular complications: T2DM without microvascular complications
  Interventions: Procedure: Blood sample collection

INTERVENTIONS:
Procedure: Blood sample collection — Collection of blood sample

SUMMARY:
Adults with diabetes mellitus have 2-3 times fold increased cardiovascular (CV) risk compared to adults without diabetes, and the risk rises with the worsening of glycaemic control. Adults with type 2 diabetes mellitus (T2DM) and microvascular complications (DMCs) have a higher risk of CV complications than subjects without DMCs. 2023 European Society of Cardiology (ESC) guidelines stated that individuals with T2DM with target organ damage (TOD), defined as presence of microvascular disease in at least three different sites (e.g., microalbuminuria (stage A2) plus retinopathy plus neuropathy), should be considered into a very high CV risk category.

Coronary artery calcium score (CACS) is a measure of the amount of calcium deposits in the coronary arteries obtained through a CT coronary imaging. CACS has become a widely available and accurate tool for determining the risk of major CV events.

The specific role of DMCs in determining the features of coronary plaques is not completely known. A recent study showed how T2DM subjects with obstructive coronary artery disease (CAD) with DMCs at their first coronary event present a more "stable" coronary atherosclerosis features at OCT-imaging, as they have a higher prevalence of fibrous plaques and healed plaques with larger calcifications compared to those with T2DM and no DMCs. In this study only subjects with obstructive CAD (defined as a stenosis ≥50% in the left main coronary artery or any stenosis ≥70% or fractional flow reserve <0.80 in any other major epicardial vessel) were enrolled.

Therefore, further research to evaluate differences in CACS in T2DM subjects with no previous history of CAD with and without DMCs is required.

Aim of our study was to evaluate the presence of differences in the distribution and tomographic features of coronary plaques in T2DM subjects with no previous history of CAD with at least one DMCs, focusing on the degree of plaque calcification calculated by the CACS.

DETAILED DESCRIPTION:
Subjects with T2DM who performed CT coronary imaging, as per clinical routine practice.

They will be, therefore, divided into two groups:

* Group A: subjects with T2DM with at least one DMC, as defined:

  • Retinopathy, defined as any diabetes related eye disease (macular oedema, severe non proliferative diabetic retinopathy, proliferative diabetic retinopathy) or previous history of retinal photocoagulation therapy and/or intravitreal injections of anti- vascular endothelial growth factor (VEGF) agents.
  * Neuropathy, including any diabetes-related neurological complication (diabetic peripheral neuropathy, diabetic autonomic neuropathy).
  * Nephropathy, defined as the presence of albuminuria (urinary albumin > 30 mg/g creatinine) and/or an estimated glomerular filtration rate < 60 mL/min/1.73 m2
* Group B: subjects with T2DM without DMCs.

Following data will be collected Anthropometric parameters

* Sex
* Year of birth
* Height, expressed in m
* Weight, expressed in Kg
* BMI, calculated as weight divided by height squared

Vital signs

* Blood pressure, expressed in mmHg;
* Heart rate, expressed in bpm;
* VFA (Visceral fat area - cm2);
* SFA (subcutaneous fat area - cm2).

Medical history

* Date of diagnosis of diabetes, at least the year;
* Comorbidities;
* Year of diagnosis of comorbidities.
* Smoking habits, defined as "current smoker", "former smoker", "never smoked"

Medications

* Diabetes medications;
* Dose of each diabetes medications;
* Year of start for each diabetes medications;
* Concomitant medications;
* Dose of each concomitant medications;
* Year of start for each concomitant medication.

Cardiovascular risk scores

• SCORE2-Diabetes [12]

Blood Tests data collection

* HbA1c
* Serum Creatinine
* Total Cholesterol
* LDL Cholesterol
* HDL Cholesterol
* Triglycerides
* Transaminases
* Microalbuminuria

Blood sample collection • CRP

Cardiovascular Autonomic Tests

Following Cardiovascular autonomic tests will be performed:

* Deep breathing: The patient sits quietly and breathes deeply at six breaths a minute (five seconds in and five seconds out) for one minute. An electrocardiogram is recorded throughout the period of deep breathing, with a marker used to indicate the onset of each inspiration and expiration.
* Valsalva manoeuvre: The test is performed by the patient blowing into a mouth- piece connected to an aneroid manometer or a modified sphygmomanometer and holding it at a pressure of 40 mm Hg for 15 seconds while a continuous electrocardiogram is recorded. The manoeuvre is performed three times with one- minute intervals between.
* Lying to standing: The test is performed by measuring the patient's blood pressure with a sphygmomanometer while he is lying down quietly and again when he stands up. The postural fall in blood pressure is taken as the difference between the systolic blood pressure lying and the systolic blood pressure standing [13].

Neuropathy evaluation

* Michigan Neuropathy Screening Instrument (MNSI-Q) questionnaire [14]
* COMPASS31 questionnaire [15]
* Diabetic Neuropathy Index (DNI) questionnaire [16]
* DN4 questionnaire [17]
* Monofilament examination

Ophthalmologic evaluation

• Non mydriatic Ocular fundus photography

Coronary CTA parameters collection

* Total EAT
* EAT of atrio_ventricular sulcus
* EAT of anterior interventricular artery, both as volume and thickness
* EAT of right coronary artery
* EAT of circumfl ex coronary artery
* EAT Volume Index (cm3/m2)
* Perivascular FAI (-30 -190 UH)
* CACS (Agatston score, Volume and mass)
* Plaque grading/stenosis (Minimum, mild, intermediate, Severe), using CAD-RADS 2.0
* Plaque characteristics non-calcific, mixed and calcific plaque, evaluating any high-risk plaque profile

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent signed before any activity related to the study
2. Age 40 - 70 years, both sexes
3. Diagnosis of T2DM ≥5 years
4. CT coronary imaging performed in 60 days before enrollment

Exclusion Criteria:

1. Previous diagnosis of type 1 diabetes, late autoimmune diabetes of the adults (LADA), diabetes secondary to pancreatitis
2. Malignant disease
3. Acute/chronic inflammatory disease
4. Severe obesity

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with T2DM who performed CT coronary imaging, as per clinical routine practice.
  They will be, therefore, divided into two groups:
  * Group A: subjects with T2DM with at least one DMC
  * Group B: subjects with T2DM without DMCs
Sampling Method: Non-Probability Sample
Enrollment: 244 (Estimated)
Dates: Start 2024-05-27 (Estimated); Primary Completion 2026-05-27 (Estimated); Study Completion 2026-05-27 (Estimated)

PRIMARY OUTCOMES:
Coronary artery calcium score | 24 months
  Differences in coronary calcium score between subjects with diabetes with and with our microvascular complications